CLINICAL TRIAL: NCT06400641
Title: CGM for Improving Blood Glucose Control in Severe Patients and the Feasibility of Automatic Drug Delivery in Combination With Insulin Pumps: A Prospective Multi-center Randomized Controlled Study
Brief Title: Study on the Feasibility of Continuous Glucose Monitoring(CGM) for Improving Blood Glucose Control in Severe Patients
Status: Recruiting | Type: Observational
Sponsor: Chinese Medical Association (Network)
Responsible Party: Sponsor
Other Study IDs: ACCURATE study
Record Dates: First submitted 2024-02-20; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-02

CONDITIONS: Continuous Glucose Monitoring
Keywords: blood glucose; insulin
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Compared to traditional blood glucose monitoring (TGM), CGM can accurately capture asymptomatic hyperglycemia and hypoglycemia events that are missed by TGM, accounting for 33% and 90% of cases, respectively. Real-time CGM provides instantaneous glucose levels and can also generate alarms for hypoglycemia and hyperglycemia based on preset glucose ranges, assisting patients in making timely adjustments to their glucose levels. Clinical studies have found that glucose control guided by real-time CGM is better, and the decrease in glycosylated hemoglobin levels is positively correlated with the frequency of CGM use. More importantly, although glucose variability can be calculated using conventional blood glucose measurements taken every four to six hours, to further assess precise changes in glucose levels, more detailed and accurate continuous data are required. In this respect, CGM has unparalleled advantages over traditional blood glucose monitoring.While the use of CGM in critically ill patients is still controversial.

DETAILED DESCRIPTION:
We conducted this clinical study to compare the effectiveness of CGM and traditional blood glucose monitoring in guiding blood glucose control in critically ill patients, and to clarify the feasibility of using CGM for critically ill patients. We also aimed to explore the possible factors that affect CGM in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Age≥ 18 years and < 80 years
* ICU stay ≤48 hours
* Expected ICU stay > 24 hours
* APACHE II score≥ 8

Exclusion Criteria:

* local infection within the sensor placement area
* Laparotomy within lower abdomen
* Participated in this study before
* In other clinical trails.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: critically ill patient
Sampling Method: Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
CGM measurement | Days within the 1st week after ICU entrance
  Test
Whole blood or fingertip blood glucose measurement | Days within the 1st week after ICU entrance
  Test
ICU stay | During the ICU stay
  Days
28-day mortality rate | 28 days after ICU entrance
  Mortality
60-day mortality rate | 60 days after ICU entrance
  Mortality
Mortality rate during ICU stay | Days from ICU entrance to ICU discharge
  Mortality

SECONDARY OUTCOMES:
Serum C-peptide | Days within the 1st week after ICU entrance
  Test
Insulin levels | Days within the 1st week after ICU entrance
  Test
Thyroid hormones and other relevant hormone levels were measured | The 1st day and the 7th day after ICU entrance
  Test

CONTACTS AND LOCATIONS:
Overall Officials: Wenkui Yu, Professor, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China